CLINICAL TRIAL: NCT03417453
Title: Eye Drop Dispensers: Safety, Efficacy and Comfort.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Asaf Achiron, PI, Wolfson Medical Center
Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Eye Drop Dispensers
Record Dates: First submitted 2018-01-07; First posted 2018-01-31 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Glaucoma; Cataract; Healthy Subjects
Keywords: normal patients; eye drops dispensers; aids; glacuoma; cataract
MeSH Terms: conditions — Glaucoma; Cataract; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Drop Dispenser TYPE Opticare (Active Comparator): subject will assess TYPE 1 dispenser
  Interventions: Device: Eye Drop Dispenser TYPE Opticare
- Eye Drop Dispenser Autodrop (Active Comparator): subject will assess Autodrop dispenser
  Interventions: Device: Eye Drop Dispenser Autodrop

INTERVENTIONS:
Device: Eye Drop Dispenser TYPE Opticare — Subject will apply normal saline eye drops to them-self with various eye drop dispensers.
  Assessment of ease of use will be conducted by questioners.
  Arms: Eye Drop Dispenser TYPE Opticare
Device: Eye Drop Dispenser Autodrop — Eye Drop Dispenser Autodrop
  Arms: Eye Drop Dispenser Autodrop

SUMMARY:
One aspect to eye drop adherence is successful instillation of the drops; however, it is well known that many patients struggle with this task. Difficulties may include aiming their drops,extending their neck, preventing excess drop leakage, avoiding contamination of the bottle tip and generating enough force to expel a drop from the bottle. Instillation aids are devices that aim to ameliorate one or more of these barriers.

Several eye drop dispensers had been developed in order to improved outcomes of eye drop instillation, including improved rates of successful administration and increased patient satisfaction compared to standard eye drop bottles.

In this study we aim to compare the eye drops various installation aids

DETAILED DESCRIPTION:
subject will evaluate 2 dispensers by questioners. efficacy and safety of each one will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* glaucoma patients

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of correct application of eye drops to the eye without missing conducted by questioners. | 5 seconds after instillation of eye drops
  assessment of correct application of eye drops to the eye without missing

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf Achiron, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided